CLINICAL TRIAL: NCT00073697
Title: Depression: The Search for Treatment-Relevant Phenotypes
Brief Title: Treatment of Depression in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Ellen Frank, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01MH065376 (NIH); R01MH065376 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Depression
Keywords: Psychotherapy; Depressive disorder; Antidepressive agents; Citalopram
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Escitalopram; Interpersonal Psychotherapy; adenylate isopentenyltransferase

ARMS (3):
- 1 (Experimental): Interpersonal Psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy
- 2 (Experimental): Escitalopram
  Interventions: Drug: Escitalopram
- 3 (Experimental): Escitalopram plus IPT
  Interventions: Other: Escitalopram plus IPT

INTERVENTIONS:
Drug: Escitalopram — Participants will receive escitalopram for a minimum of 32 weeks or approximately 8 months. Participants whose symptoms become stabilized will continue the initial treatment for another 6 months.
  Arms: 2
Behavioral: Interpersonal Psychotherapy — Participants will receive interpersonal psychotherapy (IPT) for 8 months and possibly an additional 6 months.
  Arms: 1
Other: Escitalopram plus IPT — Participants whose symptoms become stabilized will continue the initial treatment for another 6 months. Those who do not will have the second treatment added to their regimen until remission occurs.
  Arms: 3

SUMMARY:
This study will determine how certain features of depressed individuals affect their responses to depression treatment.

DETAILED DESCRIPTION:
Major depression is a serious condition that can have devastating functional consequences. Although numerous depression studies have been conducted, understanding of how best to achieve long-term recovery remains limited. This study will assess the mood, personality, pharamcokinetic and genetic characteristics of depressed participants to determine the effects of these features on treatment response.

This study will be conducted at two international treatment sites, including the University of Pittsburgh and the University of Pisa, Italy. Participants will be randomly assigned to receive either interpersonal psychotherapy (IPT) or escitalopram pharmacotherapy for a minimum of 32 weeks or approximately 8 months. Participants whose symptoms become stabilized will continue the initial treatment for another 6 months; those who do not will have the second treatment added to their regimen until remission occurs. Clinical evaluations and questionnaires will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major depression

Exclusion Criteria:

* History of manic or hypomanic episodes
* History of schizophrenia or schizoaffective disorder
* Diagnosis of anorexia nervosa or bulimia nervosa
* Current psychosis
* Drug and/or alcohol dependence or abuse within 3 months prior to study entry. Participants with episodic abuse related to mood disorders will not be excluded.
* Diagnosis of antisocial personality disorder
* Diagnosis of organic affective syndrome and uncontrolled medical illness
* Pregnancy
* Require inpatient treatment for suicidal risk or psychosis
* History of an inability to tolerate any of the study treatments
* Currently receiving treatment with an effective antidepressant

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression score | Measured at Months 8 and 14
Treatment-relevant phenotypes of depression | Measured at Months 8 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, Principal Investigator — University of Pittsburgh
Locations (2):
- Western Psychiatric Institute and Clinic - Depression Prevention Program, Pittsburgh, Pennsylvania, United States
- The University of Pisa, Pisa, Italy